CLINICAL TRIAL: NCT03810313
Title: An Eighteen-Month, Two-Arm, Randomized, Double Masked, Multicenter, Phase III Study Assessing the Efficacy and Safety of Brolucizumab Versus Aflibercept in Adult Patients With Visual Impairment Due to Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: Assessing the Efficacy and Safety of Brolucizumab Versus Aflibercept in Patients With Visual Impairment Due to Macular Edema Secondary to Central Retinal Vein Occlusion
Acronym: RAVEN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated by sponsor due to increased incidences of adverse events of special interest (intraocular inflammation including retinal vasculitis, and retinal vascular occlusion), in patients dosed every 4 weeks beyond 3 initial doses.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRTH258C2302; 2018-001788-21 (EudraCT Number)
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Central Retinal Vein Occlusion
Keywords: Visual impairment; Macular edema; Central retinal vein occlusion; CRVO; Brolucizumab; Aflibercept; Vascular endothelial growth factor; VEGF; anti-VEGF
MeSH Terms: conditions — Retinal Vein Occlusion; Vision Disorders; Macular Edema | interventions — brolucizumab; aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A masked evaluating investigator was responsible for all aspects of the study except the injections and the safety assessment following the injections. An unmasked treating investigator performed the injections and assessed patient safety following the injections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): 1 intravitreal injection every 4 weeks for a total of 6 injections, followed by 48 weeks of individual flexible treatment (IFT)
  Interventions: Drug: Brolucizumab 6 mg; Other: Sham injection
- Aflibercept 2 mg (Active Comparator): 1 intravitreal injection every 4 weeks for a total of 6 injections, followed by 48 weeks of individual flexible treatment (IFT)
  Interventions: Drug: Aflibercept 2 mg; Other: Sham injection

INTERVENTIONS:
Drug: Brolucizumab 6 mg — Solution for injection (intravitreal use)
  Other Names: RTH258; ESBA1008
  Arms: Brolucizumab 6 mg
Drug: Aflibercept 2 mg — Solution for injection (Intravitreal use)
  Other Names: EYLEA®
  Arms: Aflibercept 2 mg
Other: Sham injection — Empty sterile syringe without a needle administered as a sham injection for masking. From Week 24 to Week 72 inclusive, a sham treatment was performed to maintain subject masking in case treatment with brolucizumab or aflibercept was not deemed necessary by the investigator.

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of brolucizumab in treatment of patients with macular edema (ME) secondary to central retinal vein occlusion (CRVO).

DETAILED DESCRIPTION:
The study included Screening Period (Day -28 to Day -1), double-masked treatment period (Day 1 to Week 72), and post-treatment follow-up period (Week 72 to Week 76). Treatment visits were scheduled in 4-week intervals. After 6 initial monthly injections of brolucizumab or aflibercept (loading phase), subjects entered a one-year individualized flexible treatment (IFT) phase. During the IFT phase, an assessment of disease stability was performed at each monthly visit and subjects received either an active or a sham injection. Treatment with active was interrupted when disease stability was reached.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Patients with visual impairment due to ME secondary to CRVO diagnosed < 6 months prior to screening.
* BCVA score between 78 and 23 letters, inclusive, using ETDRS visual acuity testing charts (approximate Snellen equivalent of 20/32 to 20/320) at both screening and baseline visits.

Exclusion criteria

* Concomitant conditions or ocular disorders in the study eye at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the first 12-month study period (e.g. structural damage of the fovea, vitreous hemorrhage, retinal vascular occlusion other than CRVO, retinal detachment, macular hole, or choroidal neovascularization of any cause, diabetic retinopathy (except mild non-proliferative) and diabetic macular edema).
* Any active intraocular or periocular infection or active intraocular inflammation (e.g. infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in study eye at screening or baseline
* Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 mmHg on medication, or according to investigator's judgment, at screening or baseline
* Presence of amblyopia, amaurosis or ocular disorders in the fellow eye with BCVA < 20/200 at screening (except when due to conditions whose surgery may improve VA, e.g. cataract)
* Previous treatment with any anti-VEGF therapy or investigational drugs in the study eye at any time prior to baseline
* Previous use of intraocular or periocular steroids in study eye at any time prior to baseline
* Macular laser photocoagulation (focal/grid) in the study eye at any time prior to baseline and peripheral laser photocoagulation in the study eye within 3 months prior to the baseline
* Intraocular surgery in the study eye during the 3-month period prior to baseline
* Vitreoretinal surgery in the study eye at any time prior to baseline
* Aphakia with the absence of posterior capsule in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (109):
- United States (27):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Mountain View, California
  - Novartis Investigative Site, Santa Barbara, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, New Albany, Indiana
  - Novartis Investigative Site, Leawood, Kansas
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Stoneham, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Bloomfield, New Jersey
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Monroeville, Pennsylvania
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Abilene, Texas
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Bellaire, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Madison, Wisconsin
- Australia (7):
  - Novartis Investigative Site, Albury, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Strathfield, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Canada (4):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Québec
- China (11):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- Czechia (3):
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Prague
- France (4):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (10):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
- Greece (2):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Larissa, GR
- Hungary (4):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (2):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Milan, MI
- Japan (9):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Taito-ku, Tokyo
- Malaysia (2):
  - Novartis Investigative Site, Batu Caves, Selangor
  - Novartis Investigative Site, Shah Alam, Selangor
- Novartis Investigative Site, Tilburg, Netherlands
- Novartis Investigative Site, Arecibo, Puerto Rico
- Russia (4):
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Spain (5):
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Novartis Investigative Site, Ankara, Turkey (Türkiye)
- United Kingdom (5):
  - Novartis Investigative Site, Bury Saint Edmonds, Suffolk
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Results for CRTH258C2302 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17958
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 132 sites in 19 countries
Pre-assignment Details: The study comprised a screening period of 28 days
Period: Overall Study
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Started | 247 | 246
Completed | 66 | 70
Not Completed | 181 | 176
Not completed — Study terminated by sponsor | 164 | 159
Not completed — Subject decision | 10 | 11
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Death | 2 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 247 | 246 | 493
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (13.69) | 65.2 (12.66) | 64.1 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 96 | 192
  Male | 151 | 150 | 301
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 176 | 178 | 354
  Black or African American | 7 | 8 | 15
  Asian | 62 | 58 | 120
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  American Indian or Alaska Native | 0 | 1 | 1
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) at Week 24
Description: BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance of 4 meters.
  Min and max possible scores are 0-100 letters read respectively. A higher score represents better visual functioning.
  Missing and censored BCVA values were imputed by Last observation carried forward (LOCF) as the primary approach. Observed values from both scheduled and unscheduled post-baseline visits were used for the LOCF imputation. For subjects with no post-baseline BCVA value, the baseline value was carried forward.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one Intravitreal injection of the study treatment.
Measure: Least Squares Mean (Standard Error); unit: Letters read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Letters read | 13.2 (0.85) | 16.0 (0.85)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — Non-inferiority was considered to be established if the lower limit of the corresponding 95% CI for the estimated between group difference (brolucizumab vs. aflibercept) on change from baseline in BCVA at Week 24 is > -4 letters; p = 0.173, ANOVA; Least Square Mean Difference = -2.9, 95% CI 2-sided [-5.2 to -0.5], Standard Error of Mean 1.20

2. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 40 to Week 52
Description: An average BCVA over week 40 to week 52 was calculated. BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance of 4 meters.
  Min and max possible scores are 0-100 letters read respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Week 40 to Week 52
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment.
  The number analyzed per row is the number of subjects from the FAS who had a valid assessment for both baseline and the corresponding post baseline period.
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 120 | 120
Letters read | 13.4 (15.73) | 15.4 (13.96)

3. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 64 to Week 76
Description: An average BCVA over week 64 to week 76 was calculated. BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance of 4 meters.
  Min and max possible scores are 0-100 letters read respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Week 64 to Week 76
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 109 | 113
Letters read | 14.0 (16.39) | 16.9 (13.60)

4. Secondary Outcome: Change From Baseline in BCVA by Visit up to Week 76
Description: BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance of 4 meters. Min and max possible scores are 0-100 letters read respectively. A higher score represents better visual functioning.
Time Frame: Baseline and every 4 weeks from baseline up to Week 76
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment.
  The number analyzed per row is the number of subjects from the FAS who had a valid assessment for both baseline and the corresponding post baseline visit.
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Letters read
  Week 4: number analyzed (Participants) | 237 | 236
  Week 4 | 11.3 (12.30) | 12.8 (11.00)
  Week 8: number analyzed (Participants) | 212 | 212
  Week 8 | 13.6 (13.77) | 15.0 (11.78)
  Week 12: number analyzed (Participants) | 195 | 194
  Week 12 | 14.1 (14.17) | 16.3 (12.78)
  Week 16: number analyzed (Participants) | 174 | 171
  Week 16 | 13.3 (15.37) | 17.4 (13.54)
  Week 20: number analyzed (Participants) | 164 | 156
  Week 20 | 13.9 (14.17) | 17.6 (14.68)
  Week 24: number analyzed (Participants) | 149 | 144
  Week 24 | 13.6 (14.69) | 18.1 (13.83)
  Week 28: number analyzed (Participants) | 138 | 133
  Week 28 | 12.7 (15.52) | 16.2 (13.55)
  Week 32: number analyzed (Participants) | 130 | 123
  Week 32 | 11.5 (15.96) | 15.1 (14.58)
  Week 36: number analyzed (Participants) | 120 | 122
  Week 36 | 12.6 (17.17) | 15.3 (14.05)
  Week 40: number analyzed (Participants) | 119 | 116
  Week 40 | 13.7 (15.35) | 16.7 (12.62)
  Week 44: number analyzed (Participants) | 112 | 116
  Week 44 | 13.7 (16.59) | 15.4 (14.50)
  Week 48: number analyzed (Participants) | 113 | 111
  Week 48 | 13.5 (17.11) | 16.2 (13.14)
  Week 52: number analyzed (Participants) | 113 | 110
  Week 52 | 12.9 (18.00) | 16.3 (14.13)
  Week 56: number analyzed (Participants) | 107 | 111
  Week 56 | 13.4 (16.98) | 14.9 (16.43)
  Week 60: number analyzed (Participants) | 108 | 113
  Week 60 | 13.1 (18.75) | 15.7 (13.93)
  Week 64: number analyzed (Participants) | 107 | 108
  Week 64 | 14.2 (17.06) | 17.8 (13.54)
  Week 68: number analyzed (Participants) | 93 | 101
  Week 68 | 14.2 (16.75) | 17.0 (13.88)
  Week 72: number analyzed (Participants) | 76 | 81
  Week 72 | 15.8 (14.55) | 15.2 (15.09)
  Week 76: number analyzed (Participants) | 64 | 70
  Week 76 | 17.2 (13.46) | 14.9 (13.76)

5. Secondary Outcome: Proportion of Participants With a Gain ≥ 5, 10 and 15 Letters in BCVA by Visit Compared to Baseline
Description: The summary by visit was conducted based on the BCVA observed from each of the corresponding visits.
  BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance of 4 meters.
  Min and max possible scores are 0-100 letters read respectively. A higher score represents better visual functioning.
  Every 5 letters represents 1 line of vision on the reading chart.
Time Frame: Baseline and every 4 weeks from baseline up to Week 76
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Participants
  Week 4; BCVA gain from baseline >=5: number analyzed (Participants) | 237 | 236
  Week 4; BCVA gain from baseline >=5 | 181 | 189
  Week 4; BCVA gain from baseline >=10: number analyzed (Participants) | 237 | 236
  Week 4; BCVA gain from baseline >=10 | 138 | 132
  Week 4; BCVA gain from baseline >=15: number analyzed (Participants) | 237 | 236
  Week 4; BCVA gain from baseline >=15 | 92 | 86
  Week 8; BCVA gain from baseline >=5: number analyzed (Participants) | 212 | 212
  Week 8; BCVA gain from baseline >=5 | 177 | 183
  Week 8; BCVA gain from baseline >=10: number analyzed (Participants) | 212 | 212
  Week 8; BCVA gain from baseline >=10 | 143 | 151
  Week 8; BCVA gain from baseline >=15: number analyzed (Participants) | 212 | 212
  Week 8; BCVA gain from baseline >=15 | 103 | 95
  Week 12; BCVA gain from baseline >=5: number analyzed (Participants) | 195 | 194
  Week 12; BCVA gain from baseline >=5 | 161 | 164
  Week 12; BCVA gain from baseline >=10: number analyzed (Participants) | 195 | 194
  Week 12; BCVA gain from baseline >=10 | 134 | 141
  Week 12; BCVA gain from baseline >=15: number analyzed (Participants) | 195 | 194
  Week 12; BCVA gain from baseline >=15 | 101 | 109
  Week 16; BCVA gain from baseline >=5: number analyzed (Participants) | 174 | 171
  Week 16; BCVA gain from baseline >=5 | 144 | 152
  Week 16; BCVA gain from baseline >=10: number analyzed (Participants) | 174 | 171
  Week 16; BCVA gain from baseline >=10 | 121 | 134
  Week 16; BCVA gain from baseline >=15: number analyzed (Participants) | 174 | 171
  Week 16; BCVA gain from baseline >=15 | 91 | 104
  Week 20; BCVA gain from baseline >=5: number analyzed (Participants) | 164 | 156
  Week 20; BCVA gain from baseline >=5 | 135 | 136
  Week 20; BCVA gain from baseline >=10: number analyzed (Participants) | 164 | 156
  Week 20; BCVA gain from baseline >=10 | 114 | 122
  Week 20; BCVA gain from baseline >=15: number analyzed (Participants) | 164 | 156
  Week 20; BCVA gain from baseline >=15 | 83 | 101
  Week 24; BCVA gain from baseline >=5: number analyzed (Participants) | 149 | 144
  Week 24; BCVA gain from baseline >=5 | 125 | 130
  Week 24; BCVA gain from baseline >=10: number analyzed (Participants) | 149 | 144
  Week 24; BCVA gain from baseline >=10 | 101 | 115
  Week 24; BCVA gain from baseline >=15: number analyzed (Participants) | 149 | 144
  Week 24; BCVA gain from baseline >=15 | 78 | 97
  Week 28; BCVA gain from baseline >=5: number analyzed (Participants) | 138 | 133
  Week 28; BCVA gain from baseline >=5 | 112 | 116
  Week 28; BCVA gain from baseline >=10: number analyzed (Participants) | 138 | 133
  Week 28; BCVA gain from baseline >=10 | 91 | 104
  Week 28; BCVA gain from baseline >=15: number analyzed (Participants) | 138 | 133
  Week 28; BCVA gain from baseline >=15 | 69 | 83
  Week 32; BCVA gain from baseline >=5: number analyzed (Participants) | 130 | 123
  Week 32; BCVA gain from baseline >=5 | 100 | 100
  Week 32; BCVA gain from baseline >=10: number analyzed (Participants) | 130 | 123
  Week 32; BCVA gain from baseline >=10 | 78 | 89
  Week 32; BCVA gain from baseline >=15: number analyzed (Participants) | 130 | 123
  Week 32; BCVA gain from baseline >=15 | 58 | 76
  Week 36; BCVA gain from baseline >=5: number analyzed (Participants) | 120 | 122
  Week 36; BCVA gain from baseline >=5 | 101 | 104
  Week 36; BCVA gain from baseline >=10: number analyzed (Participants) | 120 | 122
  Week 36; BCVA gain from baseline >=10 | 86 | 84
  Week 36; BCVA gain from baseline >=15: number analyzed (Participants) | 120 | 122
  Week 36; BCVA gain from baseline >=15 | 61 | 69
  Week 40; BCVA gain from baseline >=5: number analyzed (Participants) | 119 | 116
  Week 40; BCVA gain from baseline >=5 | 101 | 98
  Week 40; BCVA gain from baseline >=10: number analyzed (Participants) | 119 | 116
  Week 40; BCVA gain from baseline >=10 | 85 | 85
  Week 40; BCVA gain from baseline >=15: number analyzed (Participants) | 119 | 116
  Week 40; BCVA gain from baseline >=15 | 59 | 71
  Week 44; BCVA gain from baseline >=5: number analyzed (Participants) | 112 | 116
  Week 44; BCVA gain from baseline >=5 | 89 | 99
  Week 44; BCVA gain from baseline >=10: number analyzed (Participants) | 112 | 116
  Week 44; BCVA gain from baseline >=10 | 75 | 82
  Week 44; BCVA gain from baseline >=15: number analyzed (Participants) | 112 | 116
  Week 44; BCVA gain from baseline >=15 | 59 | 67
  Week 48; BCVA gain from baseline >=5: number analyzed (Participants) | 113 | 111
  Week 48; BCVA gain from baseline >=5 | 92 | 89
  Week 48; BCVA gain from baseline >=10: number analyzed (Participants) | 113 | 111
  Week 48; BCVA gain from baseline >=10 | 72 | 79
  Week 48; BCVA gain from baseline >=15: number analyzed (Participants) | 113 | 111
  Week 48; BCVA gain from baseline >=15 | 56 | 63
  Week 52; BCVA gain from baseline >=5: number analyzed (Participants) | 113 | 110
  Week 52; BCVA gain from baseline >=5 | 89 | 92
  Week 52; BCVA gain from baseline >=10: number analyzed (Participants) | 113 | 110
  Week 52; BCVA gain from baseline >=10 | 71 | 81
  Week 52; BCVA gain from baseline >=15: number analyzed (Participants) | 113 | 110
  Week 52; BCVA gain from baseline >=15 | 58 | 67
  Week 56; BCVA gain from baseline >=5: number analyzed (Participants) | 107 | 111
  Week 56; BCVA gain from baseline >=5 | 88 | 92
  Week 56; BCVA gain from baseline >=10: number analyzed (Participants) | 107 | 111
  Week 56; BCVA gain from baseline >=10 | 70 | 82
  Week 56; BCVA gain from baseline >=15: number analyzed (Participants) | 107 | 111
  Week 56; BCVA gain from baseline >=15 | 58 | 64
  Week 60; BCVA gain from baseline >=5: number analyzed (Participants) | 108 | 113
  Week 60; BCVA gain from baseline >=5 | 88 | 91
  Week 60; BCVA gain from baseline >=10: number analyzed (Participants) | 108 | 113
  Week 60; BCVA gain from baseline >=10 | 72 | 80
  Week 60; BCVA gain from baseline >=15: number analyzed (Participants) | 108 | 113
  Week 60; BCVA gain from baseline >=15 | 60 | 69
  Week 64; BCVA gain from baseline >=5: number analyzed (Participants) | 107 | 108
  Week 64; BCVA gain from baseline >=5 | 88 | 89
  Week 64; BCVA gain from baseline >=10: number analyzed (Participants) | 107 | 108
  Week 64; BCVA gain from baseline >=10 | 73 | 81
  Week 64; BCVA gain from baseline >=15: number analyzed (Participants) | 107 | 108
  Week 64; BCVA gain from baseline >=15 | 59 | 65
  Week 68; BCVA gain from baseline >=5: number analyzed (Participants) | 93 | 101
  Week 68; BCVA gain from baseline >=5 | 76 | 84
  Week 68; BCVA gain from baseline >=10: number analyzed (Participants) | 93 | 101
  Week 68; BCVA gain from baseline >=10 | 61 | 72
  Week 68; BCVA gain from baseline >=15: number analyzed (Participants) | 93 | 101
  Week 68; BCVA gain from baseline >=15 | 52 | 62
  Week 72; BCVA gain from baseline >=5: number analyzed (Participants) | 76 | 81
  Week 72; BCVA gain from baseline >=5 | 65 | 63
  Week 72; BCVA gain from baseline >=10: number analyzed (Participants) | 76 | 81
  Week 72; BCVA gain from baseline >=10 | 53 | 60
  Week 72; BCVA gain from baseline >=15: number analyzed (Participants) | 76 | 81
  Week 72; BCVA gain from baseline >=15 | 46 | 50
  Week 76; BCVA gain from baseline >=5: number analyzed (Participants) | 64 | 70
  Week 76; BCVA gain from baseline >=5 | 54 | 56
  Week 76; BCVA gain from baseline >=10: number analyzed (Participants) | 64 | 70
  Week 76; BCVA gain from baseline >=10 | 47 | 49
  Week 76; BCVA gain from baseline >=15: number analyzed (Participants) | 64 | 70
  Week 76; BCVA gain from baseline >=15 | 36 | 41

6. Secondary Outcome: Proportion of Participants With a Loss ≥ 5, 10 and 15 Letters in BCVA by Visit Compared to Baseline
Description: The summary by visit was conducted based on the BCVA observed from each of the corresponding visit.
  BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance of 4 meters.
  Min and max possible scores are 0-100 letters read respectively. A higher score represents better visual functioning.
  Every 5 letters represents 1 line of vision on the reading chart.
Time Frame: Baseline and every 4 weeks from baseline up to Week 76
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Participants
  Week 4; BCVA loss from baseline >=5: number analyzed (Participants) | 237 | 236
  Week 4; BCVA loss from baseline >=5 | 10 | 7
  Week 4; BCVA loss from baseline >=10: number analyzed (Participants) | 237 | 236
  Week 4; BCVA loss from baseline >=10 | 8 | 3
  Week 4; BCVA loss from baseline >=15: number analyzed (Participants) | 237 | 236
  Week 4; BCVA loss from baseline >=15 | 5 | 2
  Week 8; BCVA loss from baseline >=5: number analyzed (Participants) | 212 | 212
  Week 8; BCVA loss from baseline >=5 | 9 | 6
  Week 8; BCVA loss from baseline >=10: number analyzed (Participants) | 212 | 212
  Week 8; BCVA loss from baseline >=10 | 7 | 3
  Week 8; BCVA loss from baseline >=15: number analyzed (Participants) | 212 | 212
  Week 8; BCVA loss from baseline >=15 | 6 | 2
  Week 12; BCVA loss from baseline >=5: number analyzed (Participants) | 195 | 194
  Week 12; BCVA loss from baseline >=5 | 9 | 7
  Week 12; BCVA loss from baseline >=10: number analyzed (Participants) | 195 | 194
  Week 12; BCVA loss from baseline >=10 | 6 | 5
  Week 12; BCVA loss from baseline >=15: number analyzed (Participants) | 195 | 194
  Week 12; BCVA loss from baseline >=15 | 5 | 1
  Week 16; BCVA loss from baseline >=5: number analyzed (Participants) | 174 | 171
  Week 16; BCVA loss from baseline >=5 | 11 | 7
  Week 16; BCVA loss from baseline >=10: number analyzed (Participants) | 174 | 171
  Week 16; BCVA loss from baseline >=10 | 8 | 5
  Week 16; BCVA loss from baseline >=15: number analyzed (Participants) | 174 | 171
  Week 16; BCVA loss from baseline >=15 | 8 | 2
  Week 20; BCVA loss from baseline >=5: number analyzed (Participants) | 164 | 156
  Week 20; BCVA loss from baseline >=5 | 6 | 8
  Week 20; BCVA loss from baseline >=10: number analyzed (Participants) | 164 | 156
  Week 20; BCVA loss from baseline >=10 | 5 | 5
  Week 20; BCVA loss from baseline >=15: number analyzed (Participants) | 164 | 156
  Week 20; BCVA loss from baseline >=15 | 5 | 5
  Week 24; BCVA loss from baseline >=5: number analyzed (Participants) | 149 | 144
  Week 24; BCVA loss from baseline >=5 | 10 | 7
  Week 24; BCVA loss from baseline >=10: number analyzed (Participants) | 149 | 144
  Week 24; BCVA loss from baseline >=10 | 8 | 5
  Week 24; BCVA loss from baseline >=15: number analyzed (Participants) | 149 | 144
  Week 24; BCVA loss from baseline >=15 | 7 | 4
  Week 28; BCVA loss from baseline >=5: number analyzed (Participants) | 138 | 133
  Week 28; BCVA loss from baseline >=5 | 10 | 7
  Week 28; BCVA loss from baseline >=10: number analyzed (Participants) | 138 | 133
  Week 28; BCVA loss from baseline >=10 | 6 | 6
  Week 28; BCVA loss from baseline >=15: number analyzed (Participants) | 138 | 133
  Week 28; BCVA loss from baseline >=15 | 6 | 5
  Week 32; BCVA loss from baseline >=5: number analyzed (Participants) | 130 | 123
  Week 32; BCVA loss from baseline >=5 | 11 | 11
  Week 32; BCVA loss from baseline >=10: number analyzed (Participants) | 130 | 123
  Week 32; BCVA loss from baseline >=10 | 9 | 8
  Week 32; BCVA loss from baseline >=15: number analyzed (Participants) | 130 | 123
  Week 32; BCVA loss from baseline >=15 | 5 | 4
  Week 36; BCVA loss from baseline >=5: number analyzed (Participants) | 120 | 122
  Week 36; BCVA loss from baseline >=5 | 9 | 7
  Week 36; BCVA loss from baseline >=10: number analyzed (Participants) | 120 | 122
  Week 36; BCVA loss from baseline >=10 | 8 | 6
  Week 36; BCVA loss from baseline >=15: number analyzed (Participants) | 120 | 122
  Week 36; BCVA loss from baseline >=15 | 6 | 5
  Week 40; BCVA loss from baseline >=5: number analyzed (Participants) | 119 | 116
  Week 40; BCVA loss from baseline >=5 | 7 | 5
  Week 40; BCVA loss from baseline >=10: number analyzed (Participants) | 119 | 116
  Week 40; BCVA loss from baseline >=10 | 6 | 3
  Week 40; BCVA loss from baseline >=15: number analyzed (Participants) | 119 | 116
  Week 40; BCVA loss from baseline >=15 | 4 | 2
  Week 44; BCVA loss from baseline >=5: number analyzed (Participants) | 112 | 116
  Week 44; BCVA loss from baseline >=5 | 8 | 9
  Week 44; BCVA loss from baseline >=10: number analyzed (Participants) | 112 | 116
  Week 44; BCVA loss from baseline >=10 | 7 | 5
  Week 44; BCVA loss from baseline >=15: number analyzed (Participants) | 112 | 116
  Week 44; BCVA loss from baseline >=15 | 6 | 5
  Week 48; BCVA loss from baseline >=5: number analyzed (Participants) | 113 | 111
  Week 48; BCVA loss from baseline >=5 | 9 | 6
  Week 48; BCVA loss from baseline >=10: number analyzed (Participants) | 113 | 111
  Week 48; BCVA loss from baseline >=10 | 7 | 4
  Week 48; BCVA loss from baseline >=15: number analyzed (Participants) | 113 | 111
  Week 48; BCVA loss from baseline >=15 | 6 | 3
  Week 52; BCVA loss from baseline >=5: number analyzed (Participants) | 113 | 110
  Week 52; BCVA loss from baseline >=5 | 9 | 7
  Week 52; BCVA loss from baseline >=10: number analyzed (Participants) | 113 | 110
  Week 52; BCVA loss from baseline >=10 | 7 | 6
  Week 52; BCVA loss from baseline >=15: number analyzed (Participants) | 113 | 110
  Week 52; BCVA loss from baseline >=15 | 7 | 5
  Week 56; BCVA loss from baseline >=5: number analyzed (Participants) | 107 | 111
  Week 56; BCVA loss from baseline >=5 | 9 | 9
  Week 56; BCVA loss from baseline >=10: number analyzed (Participants) | 107 | 111
  Week 56; BCVA loss from baseline >=10 | 6 | 7
  Week 56; BCVA loss from baseline >=15: number analyzed (Participants) | 107 | 111
  Week 56; BCVA loss from baseline >=15 | 5 | 6
  Week 60; BCVA loss from baseline >=5: number analyzed (Participants) | 108 | 113
  Week 60; BCVA loss from baseline >=5 | 11 | 10
  Week 60; BCVA loss from baseline >=10: number analyzed (Participants) | 108 | 113
  Week 60; BCVA loss from baseline >=10 | 8 | 6
  Week 60; BCVA loss from baseline >=15: number analyzed (Participants) | 108 | 113
  Week 60; BCVA loss from baseline >=15 | 6 | 3
  Week 64; BCVA loss from baseline >=5: number analyzed (Participants) | 107 | 108
  Week 64; BCVA loss from baseline >=5 | 8 | 4
  Week 64; BCVA loss from baseline >=10: number analyzed (Participants) | 107 | 108
  Week 64; BCVA loss from baseline >=10 | 6 | 2
  Week 64; BCVA loss from baseline >=15: number analyzed (Participants) | 107 | 108
  Week 64; BCVA loss from baseline >=15 | 6 | 2
  Week 68; BCVA loss from baseline >=5: number analyzed (Participants) | 93 | 101
  Week 68; BCVA loss from baseline >=5 | 5 | 6
  Week 68; BCVA loss from baseline >=10: number analyzed (Participants) | 93 | 101
  Week 68; BCVA loss from baseline >=10 | 5 | 3
  Week 68; BCVA loss from baseline >=15: number analyzed (Participants) | 93 | 101
  Week 68; BCVA loss from baseline >=15 | 3 | 1
  Week 72; BCVA loss from baseline >=5: number analyzed (Participants) | 76 | 81
  Week 72; BCVA loss from baseline >=5 | 3 | 7
  Week 72; BCVA loss from baseline >=10: number analyzed (Participants) | 76 | 81
  Week 72; BCVA loss from baseline >=10 | 3 | 5
  Week 72; BCVA loss from baseline >=15: number analyzed (Participants) | 76 | 81
  Week 72; BCVA loss from baseline >=15 | 3 | 3
  Week 76; BCVA loss from baseline >=5: number analyzed (Participants) | 64 | 70
  Week 76; BCVA loss from baseline >=5 | 1 | 3
  Week 76; BCVA loss from baseline >=10: number analyzed (Participants) | 64 | 70
  Week 76; BCVA loss from baseline >=10 | 1 | 3
  Week 76; BCVA loss from baseline >=15: number analyzed (Participants) | 64 | 70
  Week 76; BCVA loss from baseline >=15 | 1 | 3

7. Secondary Outcome: Change From Baseline in CSFT Averaged Over Week 40 to Week 52
Description: Change from baseline in central subfield thickness (CSFT) averaged over Week 40 to Week 52, measured in μm by Spectral Domain Optical Coherence Tomography (SD-OCT)
Time Frame: Baseline, Week 40 to Week 52
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment. The number analyzed per row is the number of subjects from the FAS who had at least one CSFT assessment on scheduled visits over the corresponding time point
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 119 | 120
μm | -399.9 (259.22) | -434.6 (261.71)

8. Secondary Outcome: Change From Baseline in CSFT Averaged Over Week 64 to Week 76
Description: Change from baseline in central subfield thickness (CSFT) averaged over Week 64 to Week 76, measured in μm by Spectral Domain Optical Coherence Tomography (SD-OCT)
Time Frame: Baseline, Week 64 to Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 108 | 112
μm | -411.6 (259.16) | -445.7 (259.73)

9. Secondary Outcome: Change From Baseline in CSFT by Visit up to Week 76
Description: Change from baseline in central subfield thickness (CSFT) measured in μm by Spectral Domain Optical Coherence Tomography (SD-OCT)
Time Frame: Baseline, and every 4 weeks from baseline up to Week 76
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment. The number analyzed per row is the number of subjects from the FAS who had CSFT data available on baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
μm
  Week 4: number analyzed (Participants) | 235 | 235
  Week 4 | -429.5 (254.32) | -420.6 (242.68)
  Week 8: number analyzed (Participants) | 210 | 213
  Week 8 | -448.8 (265.16) | -436.1 (255.53)
  Week 12: number analyzed (Participants) | 194 | 194
  Week 12 | -468.3 (269.55) | -440.7 (251.74)
  Week 16: number analyzed (Participants) | 174 | 170
  Week 16 | -450.1 (278.67) | -470.7 (255.64)
  Week 20: number analyzed (Participants) | 163 | 156
  Week 20 | -458.1 (270.26) | -470.2 (260.46)
  Week 24: number analyzed (Participants) | 149 | 142
  Week 24 | -446.8 (274.39) | -472.4 (249.20)
  Week 28: number analyzed (Participants) | 137 | 132
  Week 28 | -383.2 (248.81) | -417.9 (269.03)
  Week 32: number analyzed (Participants) | 129 | 122
  Week 32 | -323.5 (322.95) | -395.8 (299.16)
  Week 36: number analyzed (Participants) | 116 | 122
  Week 36 | -387.8 (280.75) | -406.5 (265.67)
  Week 40: number analyzed (Participants) | 118 | 116
  Week 40 | -403.9 (269.68) | -446.6 (270.47)
  Week 44: number analyzed (Participants) | 111 | 116
  Week 44 | -404.0 (311.37) | -418.4 (271.33)
  Week 48: number analyzed (Participants) | 112 | 111
  Week 48 | -411.5 (281.09) | -457.8 (261.08)
  Week 52: number analyzed (Participants) | 112 | 110
  Week 52 | -411.3 (276.21) | -457.0 (256.40)
  Week 56: number analyzed (Participants) | 106 | 111
  Week 56 | -384.6 (313.93) | -400.8 (298.50)
  Week 60: number analyzed (Participants) | 107 | 113
  Week 60 | -396.1 (295.96) | -438.8 (254.36)
  Week 64: number analyzed (Participants) | 105 | 107
  Week 64 | -425.2 (266.66) | -462.3 (258.08)
  Week 68: number analyzed (Participants) | 91 | 99
  Week 68 | -396.3 (282.85) | -416.1 (260.79)
  Week 72: number analyzed (Participants) | 72 | 79
  Week 72 | -401.5 (276.50) | -419.0 (252.10)
  Week 76: number analyzed (Participants) | 63 | 69
  Week 76 | -421.9 (261.63) | -408.5 (251.12)

10. Secondary Outcome: Proportion of Subjects With Presence of Retinal Fluid (Intra- and/or Subretinal Fluid) in the Study Eye by Visit up to Week 76
Description: Presence of retinal fluid (intra- and/or subretinal fluid) assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Time Frame: Every 4 weeks from week 4 up to Week 76
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment. The number analyzed per row is the number of subjects from the FAS who had data at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Participants
  Week 4: number analyzed (Participants) | 236 | 235
  Week 4 | 101 | 105
  Week 8: number analyzed (Participants) | 212 | 213
  Week 8 | 54 | 68
  Week 12: number analyzed (Participants) | 195 | 194
  Week 12 | 38 | 54
  Week 16: number analyzed (Participants) | 175 | 170
  Week 16 | 37 | 43
  Week 20: number analyzed (Participants) | 164 | 156
  Week 20 | 34 | 31
  Week 24: number analyzed (Participants) | 150 | 144
  Week 24 | 26 | 30
  Week 28: number analyzed (Participants) | 138 | 133
  Week 28 | 44 | 56
  Week 32: number analyzed (Participants) | 130 | 122
  Week 32 | 63 | 55
  Week 36: number analyzed (Participants) | 120 | 122
  Week 36 | 43 | 59
  Week 40: number analyzed (Participants) | 119 | 116
  Week 40 | 32 | 40
  Week 44: number analyzed (Participants) | 112 | 116
  Week 44 | 38 | 48
  Week 48: number analyzed (Participants) | 113 | 111
  Week 48 | 36 | 40
  Week 52: number analyzed (Participants) | 113 | 110
  Week 52 | 35 | 40
  Week 56: number analyzed (Participants) | 107 | 111
  Week 56 | 42 | 48
  Week 60: number analyzed (Participants) | 108 | 113
  Week 60 | 36 | 39
  Week 64: number analyzed (Participants) | 106 | 108
  Week 64 | 29 | 41
  Week 68: number analyzed (Participants) | 93 | 100
  Week 68 | 36 | 40
  Week 72: number analyzed (Participants) | 76 | 80
  Week 72 | 25 | 27
  Week 76: number analyzed (Participants) | 64 | 70
  Week 76 | 24 | 31

11. Secondary Outcome: Proportion of Subjects With a CSFT < 300 μm for the Study Eye by Visit up to Week 76
Description: Central subfield thickness (CSFT) is measured in μm by Spectral Domain Optical Coherence Tomography (SD-OCT)
Time Frame: Every 4 weeks from week 4 up to Week 76
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment. The number analyzed per row is the number of subjects from the FAS who had non-missing CSFT assessment at the corresponding visit
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Participants
  Week 4: number analyzed (Participants) | 236 | 235
  Week 4 | 157 | 137
  Week 8: number analyzed (Participants) | 211 | 213
  Week 8 | 168 | 155
  Week 12: number analyzed (Participants) | 195 | 194
  Week 12 | 172 | 149
  Week 16: number analyzed (Participants) | 175 | 170
  Week 16 | 153 | 141
  Week 20: number analyzed (Participants) | 164 | 156
  Week 20 | 147 | 135
  Week 24: number analyzed (Participants) | 150 | 142
  Week 24 | 135 | 123
  Week 28: number analyzed (Participants) | 138 | 132
  Week 28 | 107 | 90
  Week 32: number analyzed (Participants) | 130 | 122
  Week 32 | 81 | 74
  Week 36: number analyzed (Participants) | 117 | 122
  Week 36 | 83 | 77
  Week 40: number analyzed (Participants) | 119 | 116
  Week 40 | 94 | 86
  Week 44: number analyzed (Participants) | 112 | 116
  Week 44 | 83 | 79
  Week 48: number analyzed (Participants) | 113 | 111
  Week 48 | 82 | 83
  Week 52: number analyzed (Participants) | 113 | 110
  Week 52 | 85 | 82
  Week 56: number analyzed (Participants) | 107 | 111
  Week 56 | 74 | 71
  Week 60: number analyzed (Participants) | 108 | 113
  Week 60 | 81 | 79
  Week 64: number analyzed (Participants) | 106 | 107
  Week 64 | 85 | 80
  Week 68: number analyzed (Participants) | 92 | 99
  Week 68 | 65 | 69
  Week 72: number analyzed (Participants) | 73 | 79
  Week 72 | 59 | 56
  Week 76: number analyzed (Participants) | 64 | 69
  Week 76 | 51 | 45

12. Secondary Outcome: Number of Injections Between Week 24 and Week 52 and Between Week 24 and Week 72
Description: Number of administered injections during the individualized flexible treatment (IFT) period, between Week 24 and Week 52 and between Week 24 and Week 72 are presented
Time Frame: Week 24 to Week 52 and Week 24 to Week 72
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment. The number analyzed per row is the number of subjects from the FAS who were on study treatment until week 52 and until week 72.
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 114 | 115
Injections
  Between Week 24 and Week 52 | 2.4 (1.69) | 2.6 (2.02)
  Between Week 24 and Week 72: number analyzed (Participants) | 58 | 67
  Between Week 24 and Week 72 | 4.1 (3.08) | 4.4 (3.25)

13. Secondary Outcome: Time to Recurrence After Week 20 and up to Week 76
Description: Recurrence is defined as the need for injection while showing a lack of disease stability for the first time after Week 20 and up to Week 76.
  For subjects with recurrence after the Week 20 visit, time-to-event is calculated as (first time with the lack of disease stability - the injection date on Week 20 visit + 1). For subjects without recurrence after Week 20, the censoring time will be calculated as (last visit with disease stability assessment - the injection date on Week 20 visit + 1).
Time Frame: Week 20 to Week 76
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment. The number analyzed is the number of subjects from the FAS who did not discontinue from study treatment on or before Week 20.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 160 | 163
Weeks | 12.1 [12.1 to 12.4] | 12.1 [11.4 to 13.4]

14. Secondary Outcome: Number of Subjects With Ocular and Non-ocular AEs up to Week 52 and Week 76
Description: Number of subjects with at least one ocular or non-ocular Adverse Events (AEs).
Time Frame: Baseline to Week 76
Population: Safety Analysis Set (SAF) included all subjects who received at least one intravitreal injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Participants
  Ocular AEs up to week 52 | 105 | 77
  Non-Ocular AEs up to week 52 | 103 | 107
  Ocular AEs up to week 76 | 111 | 89
  Non-Ocular AEs up to week 76 | 119 | 117

15. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (NEI VFQ-25) at Week 24, Week 52 and Week 76
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures a patient's subjective assessment of vision-related Quality of Life (QoL).
  The 11 subscales in the VFQ-25 are general vision, ocular pain, near activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. The scores on the subscales were added together for a total score, which ranged from 0 to 100. A higher score indicated better vision-related quality of life.
Time Frame: Baseline, Week 24, Week 52 and Week 76
Population: FAS-observed: The overall number of participants analyzed is the Full Analysis Set (FAS) that included all randomized subjects who received at least one intravitreal injection of the study treatment. The number analyzed per row is the number of subjects from the FAS who had NEI VFQ-25 assessment on scheduled visits.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 247 | 246
Score on a scale
  Week 24: number analyzed (Participants) | 217 | 211
  Week 24 | 5.3 (13.08) | 7.4 (12.46)
  Week 52: number analyzed (Participants) | 128 | 128
  Week 52 | 6.0 (14.83) | 9.0 (11.10)
  Week 76: number analyzed (Participants) | 104 | 111
  Week 76 | 7.4 (14.44) | 9.4 (11.66)

16. Secondary Outcome: Number of Subjects According to Their Anti-drug Antibody (ADA) Titer at Screening and Week 4, Week 12, Week 24, Week 36, Week 52 and Week 76
Description: Anti-drug antibodies (ADA) levels were assessed from subjects assigned to brolucizumab treatment only.
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 36, Week 52 and Week 76
Population: SAF-observed: Safety Analysis Set (SAF) included all subjects who received at least one intravitreal injection with brolucizumab. The number analyzed is the number of subjects from the SAF who had a value for ADA status on scheduled visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 247
Participants
  Baseline: number analyzed (Participants) | 244
  Baseline: Negative | 105
  Baseline: 40 | 23
  Baseline: 120 | 35
  Baseline: 360 | 34
  Baseline: 1080 | 29
  Baseline: 3240 | 13
  Baseline: 9720 | 4
  Baseline: 29200 | 1
  Week 4: number analyzed (Participants) | 226
  Week 4: Negative | 101
  Week 4: 40 | 26
  Week 4: 120 | 30
  Week 4: 360 | 35
  Week 4: 1080 | 21
  Week 4: 3240 | 8
  Week 4: 9720 | 5
  Week 4: 29200 | 0
  Week 12: number analyzed (Participants) | 187
  Week 12: Negative | 77
  Week 12: 40 | 15
  Week 12: 120 | 38
  Week 12: 360 | 28
  Week 12: 1080 | 12
  Week 12: 3240 | 14
  Week 12: 9720 | 3
  Week 12: 29200 | 0
  Week 24: number analyzed (Participants) | 146
  Week 24: Negative | 51
  Week 24: 40 | 16
  Week 24: 120 | 32
  Week 24: 360 | 21
  Week 24: 1080 | 15
  Week 24: 3240 | 8
  Week 24: 9720 | 3
  Week 24: 29200 | 0
  Week 36: number analyzed (Participants) | 114
  Week 36: Negative | 35
  Week 36: 40 | 8
  Week 36: 120 | 20
  Week 36: 360 | 28
  Week 36: 1080 | 11
  Week 36: 3240 | 9
  Week 36: 9720 | 3
  Week 36: 29200 | 0
  Week 52: number analyzed (Participants) | 114
  Week 52: Negative | 37
  Week 52: 40 | 15
  Week 52: 120 | 22
  Week 52: 360 | 16
  Week 52: 1080 | 14
  Week 52: 3240 | 9
  Week 52: 9720 | 1
  Week 52: 29200 | 0
  Week 76: number analyzed (Participants) | 67
  Week 76: Negative | 25
  Week 76: 40 | 8
  Week 76: 120 | 14
  Week 76: 360 | 7
  Week 76: 1080 | 7
  Week 76: 3240 | 5
  Week 76: 9720 | 1
  Week 76: 29200 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 4 weeks post treatment, up to maximum duration of 76 weeks
Description: Any sign or symptom that occurs during the study treatment plus the 4 weeks post treatment
Groups:
- Brolucizumab 6mg; Aflibercept 2mg: 1 intravitreal injection every 4 weeks for a total of 6 injections, followed by 48 weeks of individual flexible treatment (IFT)
- Overall: Overall
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg | Overall
All-Cause Mortality (participants affected / at risk) | 2/247 | 1/246 | 3/493
Serious Adverse Events (participants affected / at risk) | 36/247 | 19/246 | 55/493
Other Adverse Events (participants affected / at risk) | 104/247 | 87/246 | 191/493
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=247) | Aflibercept 2mg (N=246) | Overall (N=493)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 0 | 1
Cataract - Fellow eye (Eye disorders) | 0 | 1 | 1
Cataract - Study eye (Eye disorders) | 0 | 1 | 1
Epiretinal membrane - Fellow eye (Eye disorders) | 1 | 0 | 1
Ocular hypertension - Study eye (Eye disorders) | 1 | 0 | 1
Retinal artery occlusion - Study eye (Eye disorders) | 2 | 0 | 2
Retinal ischaemia - Study eye (Eye disorders) | 0 | 1 | 1
Retinal vasculitis - Study eye (Eye disorders) | 2 | 0 | 2
Retinal vein occlusion - Study eye (Eye disorders) | 1 | 0 | 1
Uveitis - Study eye (Eye disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 4 | 2 | 6
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 1
Dacryocystitis - Study eye (Infections and infestations) | 1 | 0 | 1
Emphysematous cystitis (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 1
Endophthalmitis - Study eye (Infections and infestations) | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Renal cyst infection (Infections and infestations) | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Aneurysm (Vascular disorders) | 2 | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=247) | Aflibercept 2mg (N=246) | Overall (N=493)
Cataract - Study eye (Eye disorders) | 8 | 4 | 12
Conjunctival haemorrhage - Study eye (Eye disorders) | 16 | 11 | 27
Dry eye - Fellow eye (Eye disorders) | 5 | 5 | 10
Dry eye - Study eye (Eye disorders) | 6 | 6 | 12
Eye pain - Study eye (Eye disorders) | 9 | 6 | 15
Glaucoma - Fellow eye (Eye disorders) | 5 | 5 | 10
Glaucoma - Study eye (Eye disorders) | 5 | 5 | 10
Macular oedema - Study eye (Eye disorders) | 18 | 11 | 29
Ocular hypertension - Study eye (Eye disorders) | 6 | 3 | 9
Retinal ischaemia - Study eye (Eye disorders) | 6 | 1 | 7
Retinal vein occlusion - Study eye (Eye disorders) | 7 | 1 | 8
Uveitis - Study eye (Eye disorders) | 8 | 0 | 8
Visual acuity reduced - Study eye (Eye disorders) | 22 | 9 | 31
Vitreous detachment - Study eye (Eye disorders) | 11 | 11 | 22
Vitreous floaters - Study eye (Eye disorders) | 5 | 11 | 16
COVID-19 (Infections and infestations) | 5 | 6 | 11
Nasopharyngitis (Infections and infestations) | 8 | 6 | 14
Tooth abscess (Infections and infestations) | 1 | 5 | 6
Urinary tract infection (Infections and infestations) | 7 | 3 | 10
Intraocular pressure increased - Study eye (Investigations) | 10 | 13 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Headache (Nervous system disorders) | 3 | 8 | 11
Hypertension (Vascular disorders) | 19 | 10 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03810313/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03810313/SAP_001.pdf